CLINICAL TRIAL: NCT04159324
Title: StroCare - Optimised Cross-sectoral, Coordinated Treatment of Stroke Patients With Patient-orientated Outcome Measurement
Brief Title: StroCare - Optimised Cross-sectoral,Coordinated Treatment of Stroke Patients With Patient-orientated Outcome Measurement
Acronym: StroCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Albertinen Krankenhaus (Other); Elbe Kliniken Stade-Buxtehude GmbH (Unknown); Reha Centrum Hamburg GmbH (Unknown); Klinikum Bad Bramstedt GmbH (Unknown); MediClin Klinikum Soltau GmbH (Unknown); VAMED Klinik Geesthacht (Unknown); VAMED Rehaklinik Damp (Unknown); BARMER Krankenkasse (Unknown); Lohmann und Birkner medizinisches ServiceCenter GmbH (Unknown); Forcare GmbH (Other)
Responsible Party: Principal Investigator, Götz Thomalla, MD, Prof. Dr, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 01NVF18022
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: Stroke; Patient-reported outcomes (PROs); Cross-sectoral care; Stroke aftercare; Aftercare coordination; Post-rehabilitation support; Evidence based treatment; Patient-centred care; Quality of life; Morbidity; Mortality; Functional status; Feasibility; Acceptance; Process evaluation; Health economics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: For a 12-months period patients undergoing aftercare treatment as usual are enrolled as an active control group. Subsequently, the intervention is implemented (StroCare treatment) and enrolment of the intervention group takes place for another 12 months. Patients in both groups are assessed after the index ischemic event and 12 months thereafter. Further sources of information are the medical record, the electronic portal (only intervention group), routine data provided by the collaborating BARMER health insurance agency (for the intervention and control group and additionally for a historic control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StroCare treatment group (Experimental): Optimized cross-sectoral, structured and coordinated treatment pathway that integrates a patient-centred outcome evaluation
  Interventions: Other: optimized cross-sectoral, structured and coordinated treatment pathway that integrates a patient-centred outcome evaluation
- control group (No Intervention): routine aftercare stroke treatment

INTERVENTIONS:
Other: optimized cross-sectoral, structured and coordinated treatment pathway that integrates a patient-centred outcome evaluation — the optimized treatment pathway includes coordinated transitions between rehabilitation phases and institutes using individual case management and portal solutions
  Arms: StroCare treatment group

SUMMARY:
The Trial is a multi-centred controlled interventional study with a pre-post design. The primary aim of the study is the evaluation of the effectiveness and cost-effectiveness of the StroCare treatment.

DETAILED DESCRIPTION:
Stroke is the second most common cause of death in Germany and the most common cause for life-long disability in adulthood. After stroke, patients often experience incisive changes in their health, daily routine and quality of life. The developed model of care (StroCare treatment) forms a cross--sectoral, structured and coordinated treatment pathway that integrates a patient-centred outcome evaluation. It aims to optimize the transition from acute inpatient treatment after an acute stroke to the ambulant neurological rehabilitation treatment. This is done firstly by creating an electronic portal solution for a safe and coordinated transmission of clinical data between the three participating hospitals and five stroke-specialized ambulant rehabilitation clinics and secondly by introducing a case-manager provided by the participating health insurance agency for patient support and aftercare coordination. The presented study is a multi-centred controlled interventional study with a pre-post design. Stroke patients in both groups are assessed after the index ischemic event and 12 months thereafter. Further sources of information are the medical record, the electronic portal (only intervention group), and routine data provided by the collaborating BARMER health insurance agency (for the Intervention and control group and additionally for a historic control). The main hypotheses are : (1) The StroCare treatment is more effective than the routine aftercare treatment (primary outcome: patient-reported physical quality of life) and (2) the StroCare treatment reduces costs for care and in the inpatient sector by providing more coordinated and thorough rehabilitation and outpatient aftercare.

ELIGIBILITY:
Inclusion Criteria:

* Patients in inpatient care in the stroke unit of one of the participating acute clinics who are insured at the BARMER health insurance agency with the following diagnosis (ICD-10):
* Ischemic attack (I63)
* Transient ischemic attack and related syndromes (G45)
* Intracerebral haermorrhage (I64)
* Written informed consent
* Sufficient mastery of German language

Exclusion Criteria:

* Substantially impaired communication capacity due to aphasia or dementia
* Patients with artificial Respiration
* Insufficient adherence
* Premorbid score of mRS≥4
* Patients with artificial Respiration (Z99.1)
* Dementia (F00.x., F01.x. or G30.x) or aphasia (R47)
* Death during inpatient Treatment or the Admission to a nursing home following the acute treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Patient-reported physical QoL: PROMIS-10 | 1 year after index ischemic event
  Patient-reported physical Quality of Life measured with Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10); one of two provided global scores: Global Physcial Health with scores ranging from 0-20 and higher scores indicating better health state.

SECONDARY OUTCOMES:
Patient-reported mental QoL | 1 year after index ischemic event
  Patient-reported mental Quality of Life measured with Patient-Reported Outcomes Measurement Information System-10 (PROMIS-10); one of two provided global scores: Global Mental Health with scores ranging from 0-20 and higher scores indicating better health state.
Patient-reported mental health status | 1 year after index ischemic event
  Patient reported mental health Status measured with the Patient health questionnaire (PHQ-4); the questionnaire provides two sub-scores measuring anxiety and depression with scores ranging from 0-6 each with higher scores indiciating more symptoms of anxiety or depression, respectively
Functional Status modified Rankin Scale questionnaire (smRSq) | 1 year after index ischemic event
  Functional Status measured with the modified Rankin Scale (mRS); the nRS ranges from 0 (no disability) to 6 (death)
Overall survival | 1 year after index ischemic event
  Overall survival measured with the ICHOM Standard set
Stroke recurrence | 1 year after index ischemic event
  Stroke recurrence measured with the ICHOM Standard set
Utilisation of health care Services | 1 year after index ischemic event
  Utilisation of health care Services extracted from the medical record and the electronic Portal (only Intervention Group), i.e., number of admissions to hospital, number of outpatient contacts, weekly hours of physiotherapy, speech therapy, occupational therapy
Patient' s waiting time between Treatment phases (Transition) to the ambulant neurological Rehabilitation Treatment) | 1 year after index ischemic event
  Waiting time extracted from the medical record and the electronic Portal (only Intervention Group)
Success in reahin target values of relevant risk factors (individually defined target values based on available guidelines): blood pressure | 1 year after index ischemic event
  Current values Blood Pressure will be extracted from the medical record and the electronic portal and compared to the individually defined target values based on current guidelines and individuall assessement of the overall patient's situation
Success in reahin target values of relevant risk factors (individually defined target values based on available guidelines): LDL-cholesterol | 1 year after index ischemic event
  Current values of LDL-cholesterol will be extracted from the medical record and the electronic portal and compared to the individually defined target values based on current guidelines and individuall assessement of the overall patient's situation
Success in reahin target values of relevant risk factors (individually defined target values based on available guidelines): HbA1c | 1 year after index ischemic event
  Current values of HbA1c will be extracted from the medical record and the electronic portal and compared to the individually defined target values based on current guidelines and individuall assessement of the overall patient's situation
Costs | 1 year after index ischemic event
  Routine data

CONTACTS AND LOCATIONS:
Overall Officials: Götz Thomalla, Prof. Dr., Principal Investigator — University Medical Centre Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schrage T, Glissmann C, Thomalla G, Rimmele DL, Schmidt H, Rosenkranz M, Boskamp S, Harter M, Kriston L. Process evaluation of a cross-sectoral, coordinated follow-up care of stroke patients: a qualitative study. Neurol Res Pract. 2025 Jan 23;7(1):4. doi: 10.1186/s42466-024-00360-1. PMID 39844272
- [Derived] Rimmele DL, Schrage T, Brettschneider C, Engels A, Gerloff C, Harter M, Rosenkranz M, Schmidt H, Kriston L, Thomalla G. Rationale and design of an interventional study of cross-sectoral, coordinated treatment of stroke patients with patient-orientated outcome measurement (StroCare). Neurol Res Pract. 2021 Feb 2;3(1):7. doi: 10.1186/s42466-021-00107-2. PMID 33526148